CLINICAL TRIAL: NCT07064252
Title: Educational Informed Consent Video in Neurosurgery: A Randomized Controlled Trial
Brief Title: Educational Informed Consent Video in Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felix C. Stengel, MD (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor-Investigator, Felix C. Stengel, MD, Principal Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0000687
Record Dates: First submitted 2025-06-23; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Informed Consent in Neurosurgery
Keywords: Informed consent; neurosurgery; Randomized controlled trial; video-assisted consent; Patient satisfaction; Patient comprehension
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video Group (Experimental): Video group receives standard informed consent plus an individualized procedure-specific educational video
  Interventions: Procedure: Educational Informed Consent Video; Procedure: Standard informed consent
- Control Group (Active Comparator): Control group receives standard informed consent, consisting of an in-person verbal consultation with the responsible neurosurgeon supplemented by written documentation and cranial models when applicable
  Interventions: Procedure: Standard informed consent

INTERVENTIONS:
Procedure: Educational Informed Consent Video — Individualized procedure-specific educational video. Videos are developed by a multidisciplinary collaboration of neurosurgeons, medical educators, and patient advocates. Each video is tailored based on location of the pathology, surgical approach, positioning, anticoagulation intake, and intraoperative adjuncts such as electrophysiology. Each video followes a standardized format covering anatomical considerations, preoperative care, the surgical procedure, and postoperative care including potential complications, expected recovery process, and post-surgery instructions.
  Arms: Video Group
Procedure: Standard informed consent — Standard informed consent, consisting of an in-person verbal consultation with the responsible neurosurgeon supplemented by written documentation and cranial models when applicable

SUMMARY:
This single-center randomized controlled trial addresses a critical gap in neurosurgical practice by evaluating the effectiveness of video-assisted informed consent compared to standard consent procedures.

DETAILED DESCRIPTION:
Importance: Informed consent in neurosurgery faces unique challenges due to procedural complexity and limited clinical time, with traditional methods often resulting in suboptimal patient comprehension.

Objective: To determine whether preoperative educational videos improve patient comprehension and satisfaction compared to standard consent procedures in neurosurgical patients.

Design: Single-center, non-blinded randomized controlled trial. Patients are randomized (1:1) using opaque envelope methods.

Setting: Department of Neurosurgery, Kantonsspital St. Gallen, Switzerland. Intervention: Video group receives individualized educational videos plus standard consent. Control group receives standard consent only. Videos coveres surgical indication, anatomy, procedural details, and risks.

Main Outcomes and Measures: Primary outcomes: patient comprehension via standardized questionnaires, satisfaction with consent process, psychological distress (Patient Health Questionnaire-4). Assessments conducted preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The study population comprises adult patients scheduled for elective neurosurgical intracranial tumor resection

Exclusion Criteria:

* Patients requiring emergency surgery
* Patients with cognitive impairments preventing informed consent
* Patients with significant language barriers impeding effective communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Comprehension | Measurement at two timepoints: - preoperative: within 24 hours after consenting - postoperative: within 72 hours after surgery
  The investigators assess patients' comprehension through standardized questionnaires developed for neurosurgical procedures. Comprehension is evaluated by dichotomized responses: patients answering all questions correctly versus those who did not.
Patient Satisfaction | Measurement at two timepoints: - preoperative: within 24 hours after consenting - postoperative: within 72 hours after surgery
  The investigators assess patients' satisfaction through standardized questionnaires developed for neurosurgical procedures. To measure satisfaction with consent and information delivery we use a visual analogue scale (0-100, higher scores indicating greater satisfaction).
Psychological Distress | Measurement at two timepoints: - preoperative: within 24 hours after consenting - postoperative: within 72 hours after surgery
  The investigators evaluate psychological distress using the Patient Health Questionnaire 4 (PHQ-4).
  The PHQ-4 (Patient Health Questionnaire-4) is a brief, self-administered questionnaire used to screen for both anxiety and depression. It combines the PHQ-2 (a 2-item depression screener) and the GAD-2 (a 2-item anxiety screener). The PHQ-4 is designed to be a quick and easy way to identify individuals who may be experiencing symptoms of anxiety or depression, prompting further evaluation if needed. Scoring: Each item is scored on a 4-point Likert scale (0-3), and the scores are summed for each subscale (GAD-2 and PHQ-2) and the overall PHQ-4.

SECONDARY OUTCOMES:
Satisfaction with hospital stay | Measurement at two timepoints: - preoperative: within 24 hours after consenting - postoperative: within 72 hours after surgery
  We measure satisfaction with the hospital stay and information delivery using a visual analogue scale (0-100, higher scores indicating greater satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, HOCH Health Ostschweiz, Kantonsspital St. Gallen, St.Gallen, Switzerland, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No